CLINICAL TRIAL: NCT00248625
Title: A Multi-center Study of the Safety and Efficacy of N-acetylcysteine in the Treatment of Acute Liver Failure in Pediatric Patients Not Caused by Acetaminophen.
Brief Title: N-acetylcysteine in Non-Acetaminophen Pediatric Acute Liver Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Robert Squires, Jr., MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB #: 0608007; U01DK072146 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Acute Liver Failure; Hepatic Encephalopathy
Keywords: acute liver failure; hepatic encephalopathy; acetaminophen toxicity; N-acetylcysteine
MeSH Terms: conditions — Liver Failure, Acute; Hepatic Encephalopathy | interventions — Acetylcysteine; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (NAC) (Active Comparator): Eligible children were adaptively allocated by age (less than 2 years of age or at least 2 years old) and hepatic encephalopathy (grade 0-1 or 2-4) to receive N-acetylcysteine (150 mg/kg/d) in 5% dextrose (D5W) infused over 24 hours for up to 7 consecutive days
  Interventions: Drug: N-acetylcysteine
- placebo (Placebo Comparator): Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and hepatic encephalopathy (grade 0-1 or 2-4) to receive 5% dextrose (D5W) infused over 24 hours for up to 7 consecutive
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — The study drug is administered as a continuous infusion at a dose of 150 mg/kg/day for up to 7 days following entry into the study. The infusion is discontinued at the time of death, liver transplant or discharge.
  Other Names: Mucomyst
  Arms: N-acetylcysteine (NAC)
Drug: Placebo — Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and hepatic encephalopathy (grade 0-1 or 2-4) to receive N-acetylcysteine (150 mg/kg/d) in 5% dextrose (D5W) and water or placebo consisting of an equal volume of D5W alone. Volumes were adjusted for small children. Study medications were infused over 24 hours for up to 7 consecutive days in a dedicated line without other medications. Treatment was stopped earlier than 7 days in the case of hospital discharge, liver transplantation, or death within 7 days of randomization.
  Other Names: dextrose in water
  Arms: placebo

SUMMARY:
We have completed patient enrollment in the the double blind, randomized, placebo-controlled trial of intravenous (IV) N-acetylcysteine (NAC) vs. placebo for the treatment of non-acetaminophen ALF. The purpose of this study is to examine the safety and efficacy of intravenous NAC in children with ALF for whom no antidote or other specific treatment is available. Inclusion in the NAC Study required enrollment in the Pediatric Acute Liver Failure (PALF) Study Registry.

DETAILED DESCRIPTION:
The Pediatric Acute Liver Failure (PALF) Study Group to identify, characterize, and develop management strategies for infants, children and adolescents who present with acute liver failure. The PALF study group includes 20 sites (17 in the United States, 2 in the United Kingdom, and 1 in Canada). The primary objective of the Pediatric Acute Liver Failure (PALF) study is to collect, maintain, analyze, and report clinical, epidemiological, and outcome data in children with ALF, including information derived from biospecimens.

Patients enrolled in the PALF study registry were able to enroll in the NAC study providing they met the additional required inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Meet entry criteria for and be enrolled in the Pediatric Acute Liver Failure prospective database.
* Able to be evaluated and initiate treatment within the first 24 hours of hospitalization
* Patients transferred from referring hospitals to the study site may be considered for enrollment, provided that no other treatment protocol has begun, and that no liver support device (BAL, extracorporeal liver assist device, transgenic pig perfusion) has been used or is contemplated.
* Use of fresh frozen plasma infusions will not disqualify patients from participation.

Exclusion Criteria:

* older than 18 years of age
* pregnancy
* ALF that is secondary to acute acetaminophen toxicity, mushroom poisoning, or a known malignancy.
* Patients who exhibit signs of cerebral herniation, have intractable arterial hypotension, require inotropic drugs, or demonstrate signs of sepsis (temperature ≥ 39.5o C or bacteremia) at the time of enrollment
* No exclusion will be made on the basis of race, ethnic group or gender.
* Criteria for inclusion of females and minorities will be those established in the NIH guidelines

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2000-01; Primary Completion 2009-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Squires, M.D., Principal Investigator — Children's Hospital of Pittsburgh, University of Pittsburgh
Locations (20):
- United States (17):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver Children's Hospital, Denver, Colorado
  - Emory University, Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University, Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia-Presbyterian, New York, New York
  - University of Cincinnati, Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - King's College Hospital (London, UK), London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Narkewicz MR, Dell Olio D, Karpen SJ, Murray KF, Schwarz K, Yazigi N, Zhang S, Belle SH, Squires RH; Pediatric Acute Liver Failure Study Group. Pattern of diagnostic evaluation for the causes of pediatric acute liver failure: an opportunity for quality improvement. J Pediatr. 2009 Dec;155(6):801-806.e1. doi: 10.1016/j.jpeds.2009.06.005. Epub 2009 Jul 29. PMID 19643443
- [Background] Rudnick DA, Dietzen DJ, Turmelle YP, Shepherd R, Zhang S, Belle SH, Squires R; Pediatric Acute Liver Failure Study Group. Serum alpha-NH-butyric acid may predict spontaneous survival in pediatric acute liver failure. Pediatr Transplant. 2009 Mar;13(2):223-30. doi: 10.1111/j.1399-3046.2008.00998.x. Epub 2008 Jul 17. PMID 18643912
- [Background] James LP, Alonso EM, Hynan LS, Hinson JA, Davern TJ, Lee WM, Squires RH; Pediatric Acute Liver Failure Study Group. Detection of acetaminophen protein adducts in children with acute liver failure of indeterminate cause. Pediatrics. 2006 Sep;118(3):e676-81. doi: 10.1542/peds.2006-0069. PMID 16950959
- [Background] Squires RH Jr, Shneider BL, Bucuvalas J, Alonso E, Sokol RJ, Narkewicz MR, Dhawan A, Rosenthal P, Rodriguez-Baez N, Murray KF, Horslen S, Martin MG, Lopez MJ, Soriano H, McGuire BM, Jonas MM, Yazigi N, Shepherd RW, Schwarz K, Lobritto S, Thomas DW, Lavine JE, Karpen S, Ng V, Kelly D, Simonds N, Hynan LS. Acute liver failure in children: the first 348 patients in the pediatric acute liver failure study group. J Pediatr. 2006 May;148(5):652-658. doi: 10.1016/j.jpeds.2005.12.051. PMID 16737880
- [Background] Alonso EM. Acute liver failure in children: the role of defects in fatty acid oxidation. Hepatology. 2005 Apr;41(4):696-9. doi: 10.1002/hep.20680. No abstract available. PMID 15789368
- [Background] Shneider BL, Rinaldo P, Emre S, Bucuvalas J, Squires R, Narkewicz M, Gondolesi G, Magid M, Morotti R, Hynan LS. Abnormal concentrations of esterified carnitine in bile: a feature of pediatric acute liver failure with poor prognosis. Hepatology. 2005 Apr;41(4):717-21. doi: 10.1002/hep.20631. PMID 15791615
- [Background] Sundaram SS, Alonso EM, Narkewicz MR, Zhang S, Squires RH; Pediatric Acute Liver Failure Study Group. Characterization and outcomes of young infants with acute liver failure. J Pediatr. 2011 Nov;159(5):813-818.e1. doi: 10.1016/j.jpeds.2011.04.016. Epub 2011 May 31. PMID 21621221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from an established registry of children with acute liver failure. Entry criteria: children <18 years, absence of a known chronic liver disease, biochemical evidence of acute liver injury, and a liver-based coagulopathy. Evidence of hepatic encephalopathy was required if the prothrombin time (PT) was between 15-19.9 seconds
Groups:
- Placebo: Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to placebo consisting of D5W alone. Volumes were adjusted for small children. Study medications were infused over 24 hours for up to 7 consecutive days in a dedicated line without other medications. Treatment was stopped earlier than 7 days in the case of hospital discharge, liver transplantation, or death within 7 days of randomization.
  Dextrose in water: Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive N-acetylcysteine (150 mg/kg/d) in 5% dextrose (D5W) and water or placebo consisting of an equal volume of D5W alone. Volumes were adjusted for small children. Study medications were infused over 24 hours for up to 7 consecutive days in a dedicated line without other medications.
- N-acetylcysteine (NAC): Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive NAC (150 mg/kg/d) in 5% dextrose (D5W) and water. Volumes were adjusted for small children. Study medications were infused over 24 hours for up to 7 consecutive days in a dedicated line without other medications. Treatment was stopped earlier than 7 days in the case of hospital discharge, LTx, or death within 7 days of randomization.
  N-acetylcysteine: The study drug is administered as a continuous infusion at a dose of 150 mg/kg/day for up to 7 days following entry into the study. The infusion is discontinued at the time of death, liver transplant or discharge.
Period: Overall Study
Arm/Group | Placebo | N-acetylcysteine (NAC)
Started | 92 | 92
Completed | 92 | 90
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who were randomized were included in the baseline analysis.
Groups:
- N-acetylcysteine (NAC): Eligible children were adaptively allocated by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive NAC (150 mg/kg/d) in 5% dextrose (D5W) infused over 24 hours for up to 7 consecutive days N-acetylcysteine: The study drug is administered as a continuous infusion at a dose of 150 mg/kg/day for up to 7 days following entry into the study.
- Placebo: Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive 5% dextrose (D5W) infused over 24 hours for up to 7 consecutive
  Dextrose in water: placebo consisting of an equal volume of D5W alone for up to 7 days following entry into the study
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine (NAC) | Placebo | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 92 | 184
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.7 [0.8 to 10.5] | 4.5 [1.0 to 9.5] | 4.1 [0.9 to 10.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 47 | 54 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 15 | 30
  White | 68 | 65 | 133
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 3 | 5
  United States | 61 | 68 | 129
  United Kingdom | 29 | 21 | 50
Coma Grade of Hepatic Encephalopathy [Number; unit: participants] — West Haven Criteria for hepatic encephalopathy (Grade 0 - IV ) is used for participants > 3 year of age. Coma grade IV indicates a participant who is comatose , with no reflexes, is decerebrate and has abnormal EEG changes with very slow delta activity. For participants less than 3 years the Whittington Scale was used. The Whittington scale does not use EEG changes and has only 3 levels, early (grades I and II), Mid (III) with somnolence, stupor, combativeness and Late (IV) for participants who are comatose with absent reflexes and decerebrate or decorticate posturing.
  participants
    0-1 | 65 | 68 | 133
    2-4 | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Spontaneous survival without transplant plus survival following transplantation
Time Frame: One year following randomization
Population: All participants who were enrolled in the study were included in the survival analysis
Measure: Number; unit: Participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 92 | 92
Participants | 68 | 76
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.19, Log Rank

2. Secondary Outcome: Spontaneous Recovery
Description: Survival without liver transplantation
Time Frame: One year following randomization
Population: All participants enrolled in study
Measure: Number; unit: participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 92 | 92
participants | 33 | 49
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.03, Log Rank

3. Secondary Outcome: Cumulative Percent Incidence of Transplantation by 1 Year
Time Frame: Within 1 year of randomization
Measure: Number; unit: percentage of participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 92 | 92
percentage of participants | 45 | 35
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.21, Pepe and Mori test of CIF difference

4. Secondary Outcome: Length of Hospital Stay
Time Frame: Randomization to hospital discharge
Population: All participants enrolled in study with hospital stay information, 2 participants (1 in each arm) did not have hospital discharge information.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 91 | 91
days | 103 [13 to 103] | 21 [9 to 103]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.053, Kruskal-Wallis

5. Secondary Outcome: Categorized Length of ICU Stay
Description: The length of ICU stay was categorized as number of days in ICU within 7 days of randomization, unless participant either died or received an LTx within this time period. Special categories were created for these cases.
Time Frame: Within 7 days of randomization
Measure: Number; unit: participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 92 | 92
participants
  0 days | 29 | 34
  1 day | 3 | 4
  2 days | 3 | 4
  3 days | 2 | 0
  4 days | 1 | 3
  5 days | 4 | 3
  6 days | 5 | 3
  7 days | 9 | 14
  underwent LTx w/i 7 days of randomization | 28 | 22
  died w/o LTx w/i 7 days of randomization | 8 | 5
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.29, Cochran-Armitage trend

6. Secondary Outcome: Number of Organ Systems Failing
Time Frame: Within 7 days of randomization
Measure: Number; unit: participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 92 | 92
participants
  0 | 44 | 46
  1 | 21 | 23
  2 | 15 | 12
  3 | 11 | 8
  4 | 1 | 3
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.74, Cochran-Armitage trend

7. Secondary Outcome: Highest Coma Grade of Hepatic Encephalopathy
Description: West Haven Criteria for hepatic encephalopathy (Grade 0 - IV ) is used for participants > 3 year of age. Coma grade IV indicates a participant who is comatose , with no reflexes, is decerebrate and has abnormal EEG changes with very slow delta activity. For participants less than 3 years the Whittington Scale was used. The Whittington scale does not use EEG changes and has only 3 levels, early (grades I and II), Mid (III) with somnolence, stupor, combativeness and Late (IV) for participants who are comatose with absent reflexes and decerebrate or decorticate posturing.
Time Frame: Within 7 days of randomization
Population: All enrolled participants where coma grade could be assessed. Four participants (two in each randomization arm) could not have coma grade assessed during the 7 days after randomization.
Measure: Number; unit: participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 90 | 90
participants
  0 | 28 | 27
  I | 16 | 21
  II | 20 | 19
  III | 15 | 17
  IV | 11 | 6
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.54, Cochran-Armitage tren

8. Secondary Outcome: Infectious Complication
Time Frame: Within 7 days of randomization
Measure: Number; unit: Participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 92 | 92
Participants | 20 | 21
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p = 0.86, Chi-squared

ADVERSE EVENTS:
Time Frame: Seven day randomization treatment period
Description: Regular investigator assessment
Groups:
- N-acetylcysteine (NAC): Eligible children were adaptively allocated by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive NAC (150 mg/kg/d) in 5% dextrose (D5W) infused over 24 hours for up to 7 consecutive days
  N-acetylcysteine: The study drug is administered as a continuous infusion at a dose of 150 mg/kg/day for up to 7 days following entry into the study. The infusion is discontinued at the time of death, liver transplant or discharge.
- Placebo: Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive 5% dextrose (D5W) infused over 24 hours for up to 7 consecutive
  Dextrose in water: Eligible children were adaptively allocated within strata defined by age (less than 2 years of age or at least 2 years old) and HE (grade 0-1 or 2-4) to receive NAC (150 mg/kg/d) in 5% dextrose (D5W) and water or placebo consisting of an equal volume of D5W alone. Volumes were adjusted for small children. Study medications were infused over 24 hours for up to 7 consecutive days in a dedicated line without other medications. Treatment was stopped earlier than 7 days in the case of hospital discharge, LTx, or death within 7 days of randomization.
Arm/Group | N-acetylcysteine (NAC) | Placebo
Serious Adverse Events (participants affected / at risk) | 5/92 | 4/92
Other Adverse Events (participants affected / at risk) | 19/92 | 16/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (NAC) (N=92) | Placebo (N=92)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Bradycardiac episode (Cardiac disorders) | 1 | 0
Hypoglycemia (Endocrine disorders) | 1 | 0
Aplastic Anemia (Blood and lymphatic system disorders) | 1 | 0
Epstein-Barr virus (Infections and infestations) | 1 | 0
Fever, chills, sinusitis (Infections and infestations) | 1 | 0
Small intestine ulcerations (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Hearing loss (Ear and labyrinth disorders) | 0 | 1
Bigeminy (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (NAC) (N=92) | Placebo (N=92)
Infection (Infections and infestations) | 11 | 8
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dilated and fixed pupils (Eye disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleepiness (General disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 1
High Fever (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No